CLINICAL TRIAL: NCT02297295
Title: Impact of Exercise Medicine on Lower Limb Amputees According to the Three Domains of the International Classification of Functioning
Brief Title: Impact of Exercise Medicine on Lower Limb Amputees According to the International Classification of Functioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EMA001; 2014/09AVR/175 (Other: StLuc)
Record Dates: First submitted 2014-07-10; First posted 2014-11-21 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Lower Limb Amputees
Keywords: Sequelae of; Amputation, Traumatic, Limb, Lower
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physiotherapy (Experimental): Comparing the patients to themselves (spontaneus evolution) before intervention.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy three times a week for 8 weeks according to a well-defined protocol

SUMMARY:
The purpose of this study is to determine whether exercise medicine in lower limb amputees has a impact on the three domains of the International Classification of Functioning of the WHO (function, activities and participation), and on quality of life.

DETAILED DESCRIPTION:
Exercise medicine in lower limb amputees has a positive impact on physical condition and on some cardiovascular aspects (first domain of ICF). But as the investigators know, there is no evidence that this improvement is connected with a significant benefit on the performance of daily live activities and social participation (second and third domains of the ICF).

The investigators want to determine benefits of exercise medicine on all of these domains.

ELIGIBILITY:
Inclusion Criteria:

* unilateral lower limb amputation
* amputees with prothesis
* after learning how to walk with the prothesis
* walking with or without technical aids

Exclusion Criteria:

* previous exercise training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in 6 minutes walk test | at -1, 0, 2 and 4 mounths

SECONDARY OUTCOMES:
Change in Timed Up and Go | at -1, 0, 2 and 4 mounths
Change in Satisfaction towards prothesis questionnaire (SAT-PRO) | at -1, 0, 2 and 4 mounths
  questionnaire
Change in Flexibility test | at -1, 0, 2 and 4 mounths
  measurement of distance between fingers and floor
Change in Isokinetic strength testing | at -1, 0, 2 and 4 mounths
Change in Prosthetic Profile of the Amputee | at -1, 0, 2 and 4 mounths

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Caty, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Service de médecine physique et réadapation des Cliniques Universitaires Saint-Luc, Brussels, Belgium